CLINICAL TRIAL: NCT02815293
Title: Topical Ophthalmic AGN-195263 for the Treatment of Evaporative Dry Eye
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 195263-009
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dry Eye Syndromes
Keywords: EDE; evaporative dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGN-195263 (Experimental)
  Interventions: Drug: AGN-195263
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AGN-195263 — 1 drop of AGN-195263 will be instilled in each eye twice daily.
  Arms: AGN-195263
Drug: Vehicle — 1 drop of AGN-195263 vehicle (placebo) will be instilled in each eye twice daily.
  Arms: Vehicle

SUMMARY:
The objectives of this study are twofold

* To evaluate the safety and efficacy of 0.1% AGN-195263 administered twice daily compared to its vehicle in patients with evaporative dry eye (EDE)
* To evaluate the systemic pharmacokinetics of 0.1% AGN-195263 administered twice daily in patients with EDE

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 years of age or older, at the screening (day -51) visit OR
* Females, who are naturally postmenopausal (permanent cessation of menstrual periods for at least 12 consecutive months) or are permanently sterilized (ie, eg, tubal occlusion, hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy) at the screening (day -51) visit
* In at least 1 eye, all of the following objective measures of evaporative dry eye (EDE) must be present at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits

  * Tear film break-up time (TBUT) ≥ 2 seconds and ≤ 7 seconds
  * Corneal sodium fluorescein staining score ≥ 1 and ≤ 4 (Oxford scheme)
  * Anesthetized Schirmer's tear test score ≥ 10 mm after 5 minutes
* At the standardization (day -21) and baseline (day 1) visits, patients must have:

  * Ocular Surface Disease Index© (OSDI) score > 12 (0 to 100 scale)
  * Overall ocular discomfort score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
  * Ocular burning score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
  * Blurred vision score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
* In at least 1 eye, a lower lid margin meibum quality global assessment score ≥ 1 at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits
* In at least 1 eye, the number of lower lid margin expressible meibomian glands must be ≥ 3 at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits
* Use of an artificial tear product or lid hygiene (ie, warm compress, lid massage, lid scrub) for the treatment of dry eye disease, EDE or meibomian gland disease within 1 year of the standardization (day -21) visit

Exclusion Criteria:

* Male patients with a history of, known, or suspected prostate cancer
* Male patients with a prostate-specific antigen (PSA) level ≥ 4 μg/L
* Female patients with a history of known or suspected breast, cervical, ovarian, or uterine cancer
* Female patient who is of child-bearing potential
* At standardization (day -21) and / or baseline (day 1) visits, a lower lid margin meibum quality global assessment score of non-expressible (NE) in either eye
* Patients who are currently or have used hormone replacement therapy or estrogen and /or progesterone based products (including herbal and nutritional supplements) within 90 days of the standardization (day -21) visit or anticipated use during the study
* Patients who are currently using or have used any androgen or anti-androgen treatment (including herbal and nutritional supplements), within 90 days of the standardization (day -21) visit or anticipated use during the study
* Patients who are currently using or have used any hair growth product within 90 days of the standardization (day -21) visit or anticipated use during the study
* Patients who are currently using or have used corticosteroids administered via any route within 30 days prior to the standardization (day -21) visit, or any anticipated use via any route of administration prior to the month 6 visit
* Patients who are currently using or have used oral or topical macrolides, tetracycline, tetracycline derivative drugs (including doxycycline and minocycline), retinoids (eg, isotretinoin), or calcineurin inhibitors (ie, RESTASIS®, Ikervis®) within 60 days of the standardization (day -21) visit, or anticipated use prior to the month 6 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (29):
- United States (29):
  - Arizona Eye Center, Chandler, Arizona
  - Clearsight, Fullerton, California
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - Montebello Medical Center, Inc., Montebello, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Centennial Eye and Cosmetic Associates, Centennial, Colorado
  - Specialty Eye Care, Parker, Colorado
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Eye Care Centers Management, Inc. dba Clayton Eye Center, Morrow, Georgia
  - Taustine Eye Center, Louisville, Kentucky
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Mercy Medical Research Institute, Springfield, Missouri
  - Ophthalmology Consultants, Ltd, St Louis, Missouri
  - Comprehensive Eye Care, Washington, Missouri
  - Cornerstone Eye Care, LLC, High Point, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Carolina Macula and Retina, Mt. Pleasant, South Carolina
  - Nashville Vision Associates, LLC, Nashville, Tennessee
  - Robert Cizik Eye Clinic, Houston, Texas
  - Houston Eye Associates, Kingwood, Texas
  - Brazosport Eye Institute, Lake Jackson, Texas
  - The Eye Clinic of Texas, an affiliate of Houston Eye Associates, League City, Texas
  - DCT- Shah Research, LLC dba Discovery Clinical Trials, Mission, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Stacy R. Smith, M.D., P.C., Salt Lake City, Utah
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 36 participants who enrolled in the study, 18 were randomized and received intervention to comprise the safety and Intent to Treat (ITT) populations
Pre-assignment Details: This study was terminated
Groups:
- AGN-195263: One drop of 0.1% AGN-195263 instilled in each eye twice daily
- Vehicle: One drop of AGN-195263 vehicle (placebo) instilled in each eye twice daily.
- Enrolled But Not Randomized: Run-In period before randomization
Period: Overall Study
Arm/Group | AGN-195263 | Vehicle | Enrolled But Not Randomized
Started | 10 | 8 | 18
Completed | 0 | 0 | 0
Not Completed | 10 | 8 | 18
Not completed — Study termination by sponsor | 10 | 7 | 0
Not completed — Participants not randomized | 0 | 0 | 18
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-195263 | Vehicle | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 10 | 8 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9 | 18
  >=65 years | 4 | 5 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 12 | 22
  Male | 3 | 5 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 6 | 9
  White | 8 | 6 | 10 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: weight (kg) / height (m)^2] — Population: Data missing for 6 out of the 18 participants in the enrolled but not randomized arm.
  weight (kg) / height (m)^2
    number analyzed (Participants) | 10 | 8 | 12 | 30
    (all) | 27.43 (4.4580376849013) | 27.3375 (4.8256961932969) | 29.6 (7.4233864689013) | 28.1225 (1.3197836926109)
Weight [Mean (Standard Deviation); unit: Kg] — Population: Data missing for 6 out of the 18 participants in the enrolled but not randomized arm.
  Kg
    number analyzed (Participants) | 10 | 8 | 12 | 30
    (all) | 73.32 (11.022504252664) | 74.3 (16.250384610833) | 82.68 (19.69071093745) | 76.76 (3.5637743007958)
Height [Mean (Standard Deviation); unit: cm] — Population: Data missing for 6 out of the 18 participants in the enrolled but not randomized arm.
  cm
    number analyzed (Participants) | 10 | 8 | 12 | 30
    (all) | 163.78 (8.5922988774833) | 165.0875 (17.14697039567) | 167.63 (9.8016438530597) | 165.499 (3.7800461794887)

OUTCOME MEASURES:

1. Primary Outcome: Overall Ocular Discomfort Score (0 to 4 Scale; 0=None, 4=Very Severe)
Description: The overall ocular discomfort will be assessed on a questionnaire using a 0 to 4 scale on which 0=none, 1=mild, 2=moderate, 3=severe and 4=very severe.
Time Frame: 6 month visit
Population: Efficacy analyses including the overall ocular discomfort score were planned for the intent-to-treat (ITT) population who are defined as all randomized patients. Ultimately, these analyses were not fully performed due to the early termination of the study and only six patients reaching the 6 month visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AGN-195263 | Vehicle
Number analyzed (Participants) | 3 | 3
Score on a scale | 1.66 (0.513) | 1.75 (0.204)

2. Secondary Outcome: Change From Baseline in Tearfilm Break Up Time (TBUT)
Description: For TBUT, the mean of 3 measurements of time in seconds will be computed at each visit for each eye. The mean value of the study eye will be used for analysis
Time Frame: Baseline (day 1) to 6 month visit
Population: Efficacy analyses including the change from baseline in Tearfilm Break Up Time (TBUT) were planned. Ultimately, these analyses were not fully performed due to the early termination of the study and only six patients reaching the 6 month visit.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | AGN-195263 | Vehicle
Number analyzed (Participants) | 3 | 3
Seconds | 3.18 (0.284) | 3.16 (0.286)

ADVERSE EVENTS:
Time Frame: Up to 223 days
Description: Adverse Events reported for randomized patients only
Arm/Group | AGN-195263 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/8
Other Adverse Events (participants affected / at risk) | 0/10 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-195263 (N=10) | Vehicle (N=8)
Laceration (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-195263 (N=10) | Vehicle (N=8)
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to study termination, the study was underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study was terminated, no data will be published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02815293/Prot_SAP_000.pdf